CLINICAL TRIAL: NCT02746185
Title: Efficacy and Safety of Oral Rivaroxaban for the Treatment of Venous Thromboembolism in Patients With Active Cancer. A Pilot Study.
Brief Title: Cancer Associated Thrombosis, a Pilot Treatment Study Using Rivaroxaban
Acronym: CASTA-DIVA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P141204
Record Dates: First submitted 2015-12-15; First posted 2016-04-21 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Neoplasm; Venous Thromboembolism
Keywords: cancer; venous thromboembolism; low-molecular weight heparin; rivaroxaban
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism | interventions — Rivaroxaban; Heparin, Low-Molecular-Weight; Dalteparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-molecular-weight heparin (Active Comparator): dalteparin, 200 IU/kg subcutaneously once daily for one month followed by 150 IU/kg subcutaneously once daily for 2 months
  Interventions: Drug: Low-molecular-weight heparin
- Rivaroxaban (Experimental): rivaroxaban, orally, 15 mg twice daily for 3 weeks followed by 20 mg once daily for 9 weeks
  Interventions: Drug: rivaroxaban

INTERVENTIONS:
Drug: rivaroxaban — rivaroxaban, 15 mg BD (Bis in die) for 3 weeks followed by 20mg OD (Omni die) for 9 weeks
  Other Names: xarelto
  Arms: Rivaroxaban
Drug: Low-molecular-weight heparin — dalteparin, 200 IU/kg OD for 4 weeks followed by 150 IU/kg OD for 8 weeks
  Other Names: dalteparin
  Arms: Low-molecular-weight heparin

SUMMARY:
The study will compare the efficacy and safety of oral rivaroxaban and subcutaneous dalteparin in patients with cancer associated thrombosis. It is designed as a non-inferiority open label randomized multicenter trial with blinded adjudication of outcome events.

DETAILED DESCRIPTION:
Patients with active cancer and symptomatic pulmonary embolism, proximal deep vein thrombosis, iliac or caval thrombosis will be randomly assigned to receive either dalteparin using the CLOT regimen or to oral rivaroxaban using the conventional dosage given in the Einstein studies. Experimental and control treatments will be given for three months. The main outcome at three month will include all symptomatic and incidentally discovered venous thromboembolic events including pulmonary embolism (either objectively confirmed and death due to pulmonary embolism), lower limb and upper limb deep vein thrombosis, iliac, caval and visceral thrombosis and any worsening of vascular obstruction which will be collected systematically at inclusion and at day 90. The safety end-points will consist of the rate of major bleedings and the composite of major and non-major but clinically significant bleedings at day 90. All outcome events will be blindly adjudicated by a central independent adjudication committee.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Social security affiliation
* Written informed consent
* Solid active cancer, high grade lymphoma or myeloma treated with Immunomodulatory drugs (IMiDs) (thalidomide or lenalidomide). Active cancer is defined as the presence of measurable disease or ongoing (or planned) chemotherapy, radiotherapy or targeted therapy at inclusion.
* Histologically or cytologically proven cancer.
* Symptomatic venous thromboembolism objectively confirmed diagnosed because of symptoms or discovered incidentally
* High-risk of recurrent Venous thromboembolism (VTE) defined by a score of 0 or ≥ 1, using the following criteria: female sex (+1), lung cancer (+1), breast cancer (-1) non metastatic tumor (-2), previous VTE (+1).

Exclusion Criteria:

* Exclusive adjuvant hormonal treatment with no measurable residual disease
* Sub-segmental isolated pulmonary embolism (PE) without associated proximal DVT
* Isolated distal deep vein thrombosis (DVT) of the legs
* Isolated upper-extremity DVT or superior vena cava thrombosis
* Isolated visceral thrombosis
* Platelet count < 50 000 G/L
* Active bleeding
* Hepatic disease associated with coagulopathy and clinically relevant bleeding risk including cirrhotic patients with Child Pugh B and C
* Hemostatic defect with contraindication to anticoagulant treatment at therapeutic dosage
* Vena cava filter at inclusion
* Fibrinolytic therapy within 3 days preceding inclusion
* Creatinine clearance < 30 ml/min according to Cockcroft-Gault formula
* Previous heparin-induced thrombocytopenia
* Anticoagulant treatment at curative dosage for more than 3 days before inclusion
* Pregnancy or lack of effective contraceptive treatment for women of childbearing age
* Treatment with both strong CYP3A4 and P-glycoprotein (PgP) inhibitors: protease inhibitors for HIV disease, systemic ketoconazole
* Treatment with a strong CYP3A4 inducer: rifampicin, carbamazepine, phenytoin.
* Life expectancy < 3 months
* Eastern Cooperative Oncology Group (ECOG) level 3 or 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Symptomatic DVT | 3 months
  Recurrent VTE during the 3-month treatment period including all symptomatic DVT (lower limbs distal and proximal DVTs, iliac and caval thrombosis, visceral thrombosis and deep vein thrombosis of the arm)
Symptomatic PE | 3 months
  Recurrent VTE during the 3-month treatment period including symptomatic PE
Unsuspected PE and DVT | 3 months
  Recurrent VTE during the 3-month treatment period including clinically unsuspected PE and DVT discovered incidentally
Worsening of pulmonary vascular or venous obstruction | 3 months
  Recurrent VTE during the 3-month treatment period including worsening of pulmonary vascular obstruction or venous obstruction on the systematic examinations performed at the end of the 3-month treatment period

SECONDARY OUTCOMES:
Major and clinically significant bleedings during the 3-month treatment period | 3 months
  Major bleeding is defined according to the International Society on Thrombosis and Haemostasis (ISTH) criteria and includes any bleeding resulting in death; symptomatic bleeding in a critical organ including intracranial, intra spinal, intraocular, retroperitoneal, intra articular and pericardial bleeding and muscle bleeding resulting in compartment syndrome; symptomatic bleeding resulting in a decrease in the hemoglobin concentration of at least 2g/dL or resulting in the transfusion of at least two packs of blood red cells.
Symptomatic recurrences of PE or DVT of the legs | 3 months
  excluding visceral thrombosis, upper extremity deep vein thrombosis and clinically unsuspected PE and DVT diagnosed incidentally
Major and non-major clinically significant bleedings at day 90 | 3 months
  Clinically significant non-major bleedings are defined as any bleeding requiring hospitalization or a medical intervention including temporary withholding of anticoagulant treatment to stop bleeding.
Mortality | 3 months

OTHER OUTCOMES:
Rivaroxaban plasma concentrations | 3 months
  Area under the plasma concentration versus time curve (AUC) determined using a liquid chromatography-tandem mass spectrometry method

CONTACTS AND LOCATIONS:
Overall Officials: Guy Meyer, MD, Principal Investigator — APHP - HEGP
Locations (15):
- France (15):
  - CHU Amiens - Medecine vasculaire (003), Amiens
  - CHU Angers - Medecin Interne (002), Angers
  - Espace Artois Santé, Arras
  - Hopital Saint Andre - Medecine vasculaire (015), Bordeaux
  - CHU Brest - Departement de medecin interne et pneumologie (008), Brest
  - CHU Le Bocage - Medecine interne 1 (014), Dijon
  - CHU Grenoble - Medecine vasculaire (007), Grenoble
  - CH Départemental La Roche sur Yon, La Roche-sur-Yon
  - Centre hospitalier Lyon Sud - Medecine interne (011), Lyon
  - CHRU de Nîmes - Pneumologie (012), Nîmes
  - HEGP - Pneumologie et soins intensifs (001), Paris
  - Institut Curie - Soins de support en Cancerologie (020), Paris
  - CHU Saint Etienne - Medecin vasculaire et therapeutique (006), Saint-Etienne
  - Hopital Saine Musse - Service de Medecine Vasculaire (010), Toulon
  - CHU Rangueil - Medecin Vasculaire (019), Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Planquette B, Bertoletti L, Charles-Nelson A, Laporte S, Grange C, Mahe I, Pernod G, Elias A, Couturaud F, Falvo N, Sevestre MA, Ray V, Burnod A, Brebion N, Roy PM, Timar-David M, Aquilanti S, Constans J, Bura-Riviere A, Brisot D, Chatellier G, Sanchez O, Meyer G, Girard P, Mismetti P; CASTA DIVA Trial Investigators. Rivaroxaban vs Dalteparin in Cancer-Associated Thromboembolism: A Randomized Trial. Chest. 2022 Mar;161(3):781-790. doi: 10.1016/j.chest.2021.09.037. Epub 2021 Oct 8. PMID 34627853
- [Derived] Riaz IB, Fuentes HE, Naqvi SAA, He H, Sipra QR, Tafur AJ, Padranos L, Wysokinski WE, Marshall AL, Vandvik PO, Montori V, Bryce AH, Liu H, Badgett RG, Murad MH, McBane RD 2nd. Direct Oral Anticoagulants Compared With Dalteparin for Treatment of Cancer-Associated Thrombosis: A Living, Interactive Systematic Review and Network Meta-analysis. Mayo Clin Proc. 2022 Feb;97(2):308-324. doi: 10.1016/j.mayocp.2020.10.041. Epub 2021 Jun 22. PMID 34172290